CLINICAL TRIAL: NCT04009005
Title: Clinically Isolated Syndrome and Relapsing-Remitting Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terry L. Wahls (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201908778
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Clinically Isolated Syndrome; Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: Comparison of the intervention arm to standard of care.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor blinded to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Participants will receive usual care from their treating neurologist
- Therapeutic Lifestyle (Experimental): Participants will be trained via videos from a three day in-person seminar that teaches the public about the use of a therapeutic diet and lifestyle to reduce multiple sclerosis related fatigue and improve quality of life.
  Interventions: Behavioral: Therapeutic diet and lifestyle

INTERVENTIONS:
Behavioral: Therapeutic diet and lifestyle — Educational videos, 1 individual support call from RD follwed by monthly support group meetings conducted via an internet based audio/ video conference platform. Patients will be trained on a low lectin modified paleolithic elimination diet; breathing meditation practice, and walking sessions to increase daily moderate to vigorous physiscal activity
  Arms: Therapeutic Lifestyle

SUMMARY:
A key question in efforts to reduce symptoms and improve quality of life for multiple sclerosis (MS) patients is whether a therapeutic lifestyle (diet, stress reduction and exercise) is inferior to disease-modifying drug treatments in terms of reducing multiple sclerosis related symptoms, improving function and quality of life. This study will prospectively assess the changes in quality of life and clinical outcomes in two cohorts of patients who are recently diagnosed with clinically isolated syndrome (CIS) or relapsing-remitting multiple sclerosis (RRMS) to begin answering that question.

The goal of this project is to compare a diet and therapeutic lifestyle only treatment usual care in the setting of newly diagnosed individuals with RRMS or CIS, which is the precursor to the development of MS. Due to the COVID 19 Pandemic, the study was redesigned from an in-person study to a virtual visit only study prior to enrolling study subjects.

DETAILED DESCRIPTION:
The goal of this project is to compare a diet and therapeutic lifestyle only treatment usual care in the setting of newly diagnosed individuals with RRMS or CIS, which is the precursor to the development of MS. The current standard of care typically includes disease-modifying drug treatment at the initial diagnosis of RRMS or CIS. Many patients are interested in adopting a therapeutic lifestyle as their initial approach to either RRMS or CIS. Some patients decline drug therapy due to high costs and or concerns about potential medication adverse events. There are no known scientific studies that have prospectively assessed outcomes for newly-diagnosed patients who decline disease-modifying drug treatment and instead utilized only a therapeutic diet and lifestyle to manage their MS-related symptoms. This study will prospectively investigate the effect of a therapeutic diet and lifestyle on quality of life, motor, cognitive and visual function, and brain structure in patients who have been trained and supported by the study team to utilize therapeutic diet and lifestyle to optimize neuronal health and those who are receiving usual care.

Our initial pilot study in the setting of progressive MS included diet and targeted supplements, stress reduction, exercise, and electrical stimulation of muscles and demonstrated significant reduction in fatigue, improvement in quality of life and improved mood and cognition. Subsequent pilot studies which utilized a diet-only intervention in the setting of RRMS demonstrated improved quality of life and improved walking and hand function.

Intervention arm:

This study will again utilize a multimodal approach, a low-lectin modified Paleolithic elimination diet, stress reduction (breathing meditation exercise) and an exercise (daily walking and three times a week body weight strengthening) program in the absence of drug disease modifying treatment and targeted supplements in the intervention arm. The control arm will receive usual care.

Supplements (intervention arm only) Participants will be asked to continue taking any dietary supplements they report at beginning of study with the exception of supplements that are similar to those they will be taking as part of the study which they will be asked to discontinue and replace with study-approved brands (2 grams of fish oil, 1000 mcg methylB12 , 400 mcg methyl folate, pyridoxine 1.5 mg and N acetylcysteine 500 mg per day, and 2000 IU vitamin D3 .

The study will use videos from a three day seminar that teaches the public how to utilize a therapeutic diet and lifestyle to improve cellular physiology which may favorably impact disease progression to educate study participants. A registered dietitian with training in motivational interviewing and health coaching will call participants to provide coaching and support to participants as they adopt the study diet, breathing meditation and exercise program and begin the study supplements. The study coordinator and or registered dietitian will moderate monthly support group video conference meetings for participants in the intervention arm. The control arm will receive a monthly text/ email providing a summary to a recently published clinical trial related to multiple sclerosis / clinically isolated syndrome patients that is not related to diet quality or use of a therapeutic diet or lifestyle.

AIMS Aim 1: To assess the non-inferiority in the change in perceived fatigue, quality of life, fatigue, mood and cognition compared to usual care over 12 months in newly-diagnosed, disease modifying drug treatment naïve RRMS or CIS patients within and between two groups. Group one will receive standard of care. Group two will receive telehealth support for improving health behaviors in the setting of newly diagnosed RRMS or CIS in which disease modifying treatment had been recommended and declined by the study participant. The pandemic had been declared prior to the first recruitment. The study was converted to virtual study with virtaul support and limited to patient reported outcomes

ELIGIBILITY:
Inclusion Criteria:

* 1) A diagnosis of clinically isolated syndrome (CIS) or relapsing-remitting multiple sclerosis (RRMS) or CIS according to the 2010 McDonald's criteria, confirmed by the treating neurologist within 12 months of completing the first study visit. and having received a recommendation to begin disease modifying treatment (DMT)2) Must consent to sharing the clinical notes from their primary care and neurology providers during the study period.3) Must reside within the lower 48 states within the United States.4) Agreement by the treating neurologist that the patient may enroll in the study.

Exclusion Criteria:

1) Moderate or severe mental impairment as measured by the Short Portable Mental Health Questionnaire. 2) Taking insulin or Coumadin® medication. 3) History of oxalate kidney stones, schizophrenia, or active diagnosis of eating disorder. 4) Greater than 12 months since initial diagnosis of RRMS or CIS and first study visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
MS 54 Quality of Life scale physical health score | change from baseline to 12 months
  Composite scores for physical health subscales
MS 54 Quality of Life scale mental health score | change from baseline to 12 months
  Composite scores for mental health subscales

SECONDARY OUTCOMES:
Fatigue Severity Score | Baseline to 12
  Questionnaire asking about fatigue
Modified Fatigue Impact Scale | Baseline to 12
  Questionnaire asking about fatigue
Perceived Deficits Questionnaire | Baseline to 12
  Questionnaire asking about mental clairty
Anxiety Score -Hospital Anxiety and Depression Survey | change from baseline to 12 months
  Survey asking about mood and daily activities. Change in anxiety score for the hospital anxiety and depression scale score based on the responses.
Depression score -Hospital Anxiety and Depression Survey | change from baseline to 12 months
  Survey asking about mood and daily activities. Change in depress score for the hospital anxiety and depression scale score based on the responses.
MS Clinical symptoms over time | baseline to 6 months
  Medical record abstraction of function and MS symptoms from progress notes, (worse, stable, improved)
MS Clinical symptoms over time | baseline to 12 months
  Medical record abstraction of function and MS symptoms from progress notes (worse, stable, improved)
MS Clinical symptoms over time | baseline to 18 months
  Medical record abstraction of function and MS symptoms from progress notes (worse, stable, improved)
MS Clinical symptoms over time | baseline to 24 months
  Medical record abstraction of function and MS symptoms from progress notes (worse, stable, improved)
Dietary intake | baseline to 12 months
  Automated 24 hour dietary intake questionnaire completed online that asks questions about beverages and foods consumed in the prior 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisht B, Darling WG, Grossmann RE, Shivapour ET, Lutgendorf SK, Snetselaar LG, Hall MJ, Zimmerman MB, Wahls TL. A multimodal intervention for patients with secondary progressive multiple sclerosis: feasibility and effect on fatigue. J Altern Complement Med. 2014 May;20(5):347-55. doi: 10.1089/acm.2013.0188. Epub 2014 Jan 29. PMID 24476345
- [Background] Wahls TL, Reese D, Kaplan D, Darling WG. Rehabilitation with neuromuscular electrical stimulation leads to functional gains in ambulation in patients with secondary progressive and primary progressive multiple sclerosis: a case series report. J Altern Complement Med. 2010 Dec;16(12):1343-9. doi: 10.1089/acm.2010.0080. PMID 21138391
- [Background] Reese D, Shivapour ET, Wahls TL, Dudley-Javoroski SD, Shields R. Neuromuscular electrical stimulation and dietary interventions to reduce oxidative stress in a secondary progressive multiple sclerosis patient leads to marked gains in function: a case report. Cases J. 2009 Aug 10;2:7601. doi: 10.4076/1757-1626-2-7601. PMID 19918474
- [Background] Bisht B, Darling WG, Shivapour ET, Lutgendorf SK, Snetselaar LG, Chenard CA, Wahls TL. Multimodal intervention improves fatigue and quality of life in subjects with progressive multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2015;5:19-35. doi: 10.2147/DNND.S76523. Epub 2015 Feb 27. PMID 30728736
- [Background] Irish AK, Erickson CM, Wahls TL, Snetselaar LG, Darling WG. Randomized control trial evaluation of a modified Paleolithic dietary intervention in the treatment of relapsing-remitting multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2017 Jan 4;7:1-18. doi: 10.2147/DNND.S116949. eCollection 2017. PMID 30050374
- [Background] Lee JE, Bisht B, Hall MJ, Rubenstein LM, Louison R, Klein DT, Wahls TL. A Multimodal, Nonpharmacologic Intervention Improves Mood and Cognitive Function in People with Multiple Sclerosis. J Am Coll Nutr. 2017 Mar-Apr;36(3):150-168. doi: 10.1080/07315724.2016.1255160. Epub 2017 Apr 10. PMID 28394724
- [Background] Wahls TL, Chenard CA, Snetselaar LG. Review of Two Popular Eating Plans within the Multiple Sclerosis Community: Low Saturated Fat and Modified Paleolithic. Nutrients. 2019 Feb 7;11(2):352. doi: 10.3390/nu11020352. PMID 30736445
- [Background] Chenard CA, Rubenstein LM, Snetselaar LG, Wahls TL. Nutrient Composition Comparison between a Modified Paleolithic Diet for Multiple Sclerosis and the Recommended Healthy U.S.-Style Eating Pattern. Nutrients. 2019 Mar 1;11(3):537. doi: 10.3390/nu11030537. PMID 30832289
- [Background] Fellows Maxwell K, Wahls T, Browne RW, Rubenstein L, Bisht B, Chenard CA, Snetselaar L, Weinstock-Guttman B, Ramanathan M. Lipid profile is associated with decreased fatigue in individuals with progressive multiple sclerosis following a diet-based intervention: Results from a pilot study. PLoS One. 2019 Jun 18;14(6):e0218075. doi: 10.1371/journal.pone.0218075. eCollection 2019. PMID 31211794
- [Derived] Saxby SM, Ehlinger MA, Brooks L, Titcomb TJ, Ten Eyck P, Rubenstein LM, Bisht B, Shemirani F, Gill C, Kamholtz J, Snetselaar LG, Wahls TL. Feasibility and assessment of self-reported dietary recalls among newly diagnosed multiple sclerosis: a quasi-experimental pilot study. Front Nutr. 2024 Oct 11;11:1369700. doi: 10.3389/fnut.2024.1369700. eCollection 2024. PMID 39464680
- [Derived] Saxby SM, Shemirani F, Crippes LJ, Ehlinger MA, Brooks L, Bisht B, Titcomb TJ, Rubenstein LM, Eyck PT, Hoth KF, Gill C, Kamholz J, Snetselaar LG, Wahls TL. Effects of a Remote Multimodal Intervention Involving Diet, Walking Program, and Breathing Exercise on Quality of Life Among Newly Diagnosed People with Multiple Sclerosis: A Quasi-Experimental Non-Inferiority Pilot Study. Degener Neurol Neuromuscul Dis. 2024 Jan 9;14:1-14. doi: 10.2147/DNND.S441738. eCollection 2024. PMID 38222092